CLINICAL TRIAL: NCT00399308
Title: An Initial Evaluation Of The Safety And Activity Of Celaderm(TM) Treatment Regimens In Healing Venous Leg Ulcers
Brief Title: Evaluation of Safety and Activity of Celaderm in Healing Venous Leg Ulcers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P001-001-B
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Leg Ulcer; Varicose Ulcer
Keywords: wound; leg; venous; chronic; wound healing
MeSH Terms: conditions — Leg Ulcer; Varicose Ulcer; Wounds and Injuries; Bronchiolitis Obliterans Syndrome | interventions — Compression Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Multi-layer compression bandaging (Profore)
  Interventions: Device: Control (compression bandaging)
- Celaderm, Bi-Weekly (Experimental): Celaderm, bi-weekly applications, up to a maximum of four applications
  Interventions: Device: Celaderm (Frozen Cultured Epidermal Allograft)
- Celaderm, Weekly (Experimental): Celaderm, applied weekly, up to a maximum of four applications
  Interventions: Device: Celaderm (Frozen Cultured Epidermal Allograft)

INTERVENTIONS:
Device: Celaderm (Frozen Cultured Epidermal Allograft) — Four biweekly applications of Celaderm plus compression therapy
  Other Names: Frozen Cultured Epidermal Allograft (CEA); Cultured Keratinocytes
  Arms: Celaderm, Bi-Weekly
Device: Celaderm (Frozen Cultured Epidermal Allograft) — Four weekly applications of Celaderm plus compression therapy
  Other Names: Frozen Cultured Epidermal Allograft (CEA); Cultured Keratinocytes
  Arms: Celaderm, Weekly
Device: Control (compression bandaging) — Multi-layer compression bandaging
  Other Names: Profore
  Arms: Control

SUMMARY:
This pilot study was designed to test the safety of Celaderm(TM) in treating venous leg ulcers and to give preliminary information about the efficacy of two different Celaderm(TM) dosing regimens.

DETAILED DESCRIPTION:
Celaderm(TM) weekly for four weeks or biweekly for four treatments combined with Profore(R) compression vs. Profore(R) compression alone.

ELIGIBILITY:
Inclusion Criteria:

* venous ulcer > 1 month and < 12 months in duration; 2 to 20 sq cm in surface area; not infected
* confirmatory venous ultrasound showing prior DVT and concurrent venous reflux
* ankle-brachial index 0.80 or greater

Exclusion Criteria:

* cutaneous malignancy
* recent treatment with corticosteroids or chemotherapeutic agents
* wound exposed bone, tendon or neurovascular structure
* wound infected and requiring antibiotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-01-31 (Actual); Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (9):
  - Dr. Robert Snyder, Tamarac, Florida
  - National Center for Limb Preservation, Niles, Illinois
  - Beth Israel Deaconess Medical Center, Division of Podiatry, Boston, Massachusetts
  - State University of New York Stony Brook, Stony Brook, New York
  - Center for Curative & Palliative Wound Care, Calvary Hospital, The Bronx, New York
  - University of North Carolina at Chapel Hill, Division of Vascular Surgery, Durham, North Carolina
  - Blair Medical Associates, Inc., Station Medical Center, Associates Wound Clinic, Altoona, Pennsylvania
  - Peripheral Vascular Associates, P.A., San Antonio, Texas
  - Dixie Regional Medical Center, Wound Care, St. George, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An enrollment of 55 patients was planned to produce an expected yield of approximately 45 evaluable patients at up to nine study centers.
Pre-assignment Details: 72 patients were consented in this study. Eighteen failed screening: eight had HbA1c > 7%; six failed wound size criteria; one was positive for HIV; one had a normal venous ultrasound; and two withdrew consent. Of the remaining 54 patients, 14 were not randomized: 11 healed > 50% during screening; one had a severe AE; and two more withdrew.
Groups:
- Group I - Weekly Celaderm: Weekly topical applications of Celaderm, up to a maximum of four (4) applications, in combination with Adaptic and Profore four-layer compression dressing
- Group II - Bi-weekly Celaderm: Bi-weekly topical applications of Celaderm, up to a maximum of four (4) applications, in combination with Adaptic and Profore four-layer compression dressing
- Group III - Control: Adaptic and Profore four-layer compression dressing
Period: Overall Study
Arm/Group | Group I - Weekly Celaderm | Group II - Bi-weekly Celaderm | Group III - Control
Started | 13 | 15 | 12
Completed | 13 | 15 | 11 (One patient withdrew: did not want to comply with study requirements)
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I - Weekly Celaderm | Group II - Bi-weekly Celaderm | Group III - Control | Total
Number analyzed (Participants) | 13 | 15 | 12 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 14 | 9 | 29
  >=65 years | 7 | 1 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.54 (12.65) | 60.40 (8.75) | 64 (12.85) | 65.28 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 9 | 4 | 16
  Male | 10 | 6 | 8 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 15 | 12 | 40

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy: Cumulative Proportion of Patients Completely Healed by the End of the Treatment Period, as Judged by the Investigator's Direct Observation.
Description: The primary efficacy observation was the proportion of wounds that achieved complete wound closure after 12 weeks of active treatment (i.e. of of Week 15 including screening/wash-in phase.)
Time Frame: 12 weeks
Population: Intent-to-Treat population (i.e. all subjects randomized to treatment)
Measure: Number; unit: participants
Arm/Group | Group I - Weekly Celaderm | Group II - Bi-weekly Celaderm | Group III - Control
Number analyzed (Participants) | 13 | 15 | 12
participants | 1 | 4 | 3

2. Secondary Outcome: Secondary Efficacy: Proportion of Patients Achieving 90% Re-epithelialization After 12 Weeks of Active Treatment.
Description: Re-epithelialization was judged by the Medical Monitor based upon computerized planimetry of serial wound photographs.
Time Frame: 12 Weeks
Population: Intent-to-Treat population
Measure: Number; unit: participants
Arm/Group | Group I - Weekly Celaderm | Group II - Bi-weekly Celaderm | Group III - Control
Number analyzed (Participants) | 13 | 15 | 12
participants | 1 | 5 | 3

3. Secondary Outcome: Secondary Efficacy: Durability of Wound Closure Through 12 Weeks After the End of the Treatment Period.
Description: The proportion of patients who had a recurrence of the study ulcer during follow-up after achieving wound closure during the active treatment period.
Time Frame: Variable - minimum of 12 weeks of follow-up.
Population: Intent-to-treat population achieving primary outcome
Measure: Number; unit: participants
Arm/Group | Group I - Weekly Celaderm | Group II - Bi-weekly Celaderm | Group III - Control
Number analyzed (Participants) | 1 | 4 | 3
participants | 0 | 1 | 0

4. Secondary Outcome: Secondary Efficacy: Cumulative Proportion of Patients Completely Healed by the End of the Follow-up Period (24 Weeks).
Description: The proportion of patients achieving wound closure by the end of the study follow-up period, 90 days after the end of the active treatment period.
Time Frame: 24 weeks
Population: Intent-to-Treat population
Measure: Number; unit: participants
Arm/Group | Group I - Weekly Celaderm | Group II - Bi-weekly Celaderm | Group III - Control
Number analyzed (Participants) | 13 | 15 | 12
participants | 3 | 7 | 5

ADVERSE EVENTS:
Arm/Group | Group I - Weekly Celaderm | Group II - Bi-weekly Celaderm | Group III - Control
Serious Adverse Events (participants affected / at risk) | 1/13 | 2/15 | 5/12
Other Adverse Events (participants affected / at risk) | 3/13 | 2/15 | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I - Weekly Celaderm (N=13) | Group II - Bi-weekly Celaderm (N=15) | Group III - Control (N=12)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — Cellulitis of the study or non-study leg
Acute Exacerbation of Chronic Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Critical Limb Ischemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Siezure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group I - Weekly Celaderm (N=13) | Group II - Bi-weekly Celaderm (N=15) | Group III - Control (N=12)
Ulcer Infection (Infections and infestations) | 3 (4) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations of the trial include the potential for outcome assessment bias as the study was not blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No